CLINICAL TRIAL: NCT01114880
Title: A Phase 3, Randomized, Double-Blind, Placebo Controlled, Multicenter, Efficacy and Safety Study of Adalimumab in Adult Chinese Subjects With Active Ankylosing Spondylitis
Brief Title: Efficacy and Safety of Adalimumab in Adult Chinese Subjects With Active Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M11-991
Record Dates: First submitted 2010-02-05; First posted 2010-05-03 (Estimated); Results first posted 2011-11-04 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis; China
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Blinded placebo from Week 0 to Week 10, open-label adalimumab from Week 12 to Week 24.
  Interventions: Biological: adalimumab; Other: placebo
- Adalimumab (Experimental): Blinded adalimumab from Week 0 to Week 10, open-label adalimumab from Week 12 to Week 24.
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — Prefilled syringe, 40 mg/0.8 mL administered subcutaneously every other week
  Other Names: ABT-D2E7; Humira
Other: placebo — Prefilled syringe, matching placebo administered subcutaneously every other week
  Arms: Placebo

SUMMARY:
Study of the efficacy and safety of adalimumab compared with placebo in adult Chinese participants with ankylosing spondylitis (AS) who have had an inadequate response to or who are intolerant to one or more nonsteroidal anti-inflammatory drugs (NSAIDs)

DETAILED DESCRIPTION:
Adults with active ankylosing spondylitis (AS) were randomized in a 2:1 ratio to receive treatment with adalimumab 40 mg every other week (eow) or matching placebo, given subcutaneously (SC), in the 12-week double-blind (DB) phase. Randomized participants received one SC injection of the appropriate DB study medication (adalimumab 40 mg or matching placebo) at Week 0 and then eow until Week 10. Participants who completed the DB phase could enter the 12-week open-label (OL) phase, during which all participants received treatment with adalimumab 40 mg eow, starting at Weeks 12 through 22. No study drug was administered or injected at the final study visit (Week 24). A follow-up visit occurred 70 days after the last dose of study drug (in DB or OL phases) to obtain information on any ongoing or new adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 65 years
* Has a diagnosis of ankylosing spondylitis (AS) based on the Modified New York Criteria
* Has active AS, as defined by fulfillment of at least 2 of the following 3 conditions at both Screening and Baseline visits:

  * BASDAI score at least 4 cm
  * Total back pain on a visual analog scale (VAS) at least 40 mm
  * Morning stiffness at least 1 hr
* Has inadequate response to or intolerance to one or more non-steroidal anti-inflammatory drugs (NSAIDs) as defined by the Investigator

Exclusion Criteria:

* Has total spinal ankylosis (bamboo spine)
* Has undergone spinal surgery or joint surgery involving joints assessed within 2 months prior to Baseline
* Has extra-articular manifestations (i.e., psoriasis, uveitis, inflammatory bowel disease) that is not clinically stable, as defined by the Investigator's best clinical judgment, for at least 28 days prior to Baseline
* Has received intra-articular joint injection(s), spinal or paraspinal injection(s) with corticosteroids within 28 days prior to Baseline
* Has prior exposure to any biologic therapy with potential therapeutic impact on AS, including anti-TNF (tumor necrosis factor) therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aileen Pangan, Study Director — Abbott
Locations (9):
- China (9):
  - Site Reference ID/Investigator# 24054, Hefei, AN
  - Site Reference ID/Investigator# 25522, Beijing
  - Site Reference ID/Investigator# 24055, Beijing
  - Site Reference ID/Investigator# 24052, Beijing
  - Site Reference ID/Investigator# 24056, Guangzhou
  - Site Reference ID/Investigator# 24243, Hangzhou
  - Site Reference ID/Investigator# 24053, Shanghai
  - Site Reference ID/Investigator# 24058, Shanghai
  - Site Reference ID/Investigator# 24057, Xi'an

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab: Blinded adalimumab from Week 0 to Week 10, open-label adalimumab from Week 12 to Week 22
- Placebo: Blinded placebo from Week 0 to Week 10, open-label adalimumab from Week 12 to Week 22
Period: Period 1 (Week 0 to Week 12)
Arm/Group | Adalimumab | Placebo
Started | 229 | 115
Completed | 224 | 113
Not Completed | 5 | 2
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Poor subject compliance | 0 | 1
Period: Period 2 (Week 12 to Week 24)
Arm/Group | Adalimumab | Placebo
Started | 224 | 113
Completed | 221 | 111
Not Completed | 3 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab | Placebo | Total
Number analyzed (Participants) | 229 | 115 | 344
Age Continuous [Mean (Standard Deviation); unit: years] | 30.1 (8.73) | 29.6 (7.49) | 29.9 (8.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 20 | 64
  Male | 185 | 95 | 280
Region of Enrollment [Number; unit: participants]
  China | 229 | 115 | 344

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Meeting the Assessment of Spondyloarthritis International Society (ASAS) ASAS20 Response Criteria
Description: ASAS20 responder had improvement of 20% or more and absolute improvement of at least 10 units (on a scale of 0 [least] to 100 [worst]) from Baseline in at least 3 of the following 4 domains, with absence of deterioration (change for worse of at least 20% and net worsening of at least 10 units) in the potential remaining domain: Patient's Global Assessment of Disease Activity; Total Back Pain visual analog scale (VAS); Bath Ankylosing Spondylitis Functional Index (BASFI); and Inflammation (mean of 2 morning stiffness-related Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] scores).
Time Frame: Week 12
Population: Analysis was performed on the Intent-to-Treat (ITT) analysis set, which included all subjects who were randomized and received at least 1 dose of double-blind study drug. A non-responder (NRI) imputation was used in which a missing response was imputed as non-response.
Measure: Number; unit: participants
Groups:
- Adalimumab/Adalimumab: Blinded adalimumab from Week 0 to Week 10; open-label adalimumab from Week 12 to Week 22
- Placebo/Adalimumab: Blinded Placebo from Week 0 to Week 10; open-label adalimumab from Week 12 to Week 22
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 229 | 115
participants | 154 | 35
Statistical Analysis 1: Comparison: Adalimumab/Adalimumab vs Placebo/Adalimumab; Test type: Superiority or Other; p < 0.001, Chi-squared

2. Secondary Outcome: Number of Participants Meeting the ASAS20 Response Criteria
Description: as for outcome 1
Time Frame: Week 24
Population: ITT analysis set, missing data imputed by NRI
Measure: Number; unit: participants
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 224 | 113
participants | 180 | 85

3. Secondary Outcome: Number of Participants Meeting the ASAS40 Response Criteria
Description: An ASAS40 responder had improvement of 40% or more and absolute improvement of 20 units or more (on a scale of 0 [least] to 100 [worst]) from Baseline in at least 3 of the 4 domains identified above for the ASAS20. In addition, there must have been an absence of deterioration in the potential remaining domain, where deterioration was defined as a net worsening of greater than 0 units (on a scale of 0 to 100).
Time Frame: Week 12
Population: ITT analysis set, missing data imputed by NRI
Measure: Number; unit: participants
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 229 | 115
participants | 102 | 11
Statistical Analysis 1: Comparison: Adalimumab/Adalimumab vs Placebo/Adalimumab; Test type: Superiority or Other; p < 0.001, Chi-squared

4. Secondary Outcome: Number of Participants Meeting the ASAS40 Response Criteria
Description: as for outcome 3
Time Frame: Week 24
Population: ITT analysis set, missing data imputed by NRI
Measure: Number; unit: participants
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 224 | 113
participants | 134 | 63

5. Secondary Outcome: Number of Participants Meeting the ASAS5/6 Response Criteria
Description: An ASAS5/6 responder had an improvement from Baseline of 20% or more in 5 of the following 6 domains: Patient's Global Assessment of Disease Activity; pain as measured by the Total Back Pain visual analog scale (VAS); function as measured by the Bath Ankylosing Spondylitis Functional Index (BASFI); inflammation (mean of 2 morning stiffness-related Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] scores); spinal mobility (lateral lumbar flexion from Bath Ankylosing Spondylitis Metrology Index [BASMI]); and acute phase reactant (high-sensitivity C-reactive protein).
Time Frame: Week 12
Population: ITT analysis set, missing data imputed by NRI
Measure: Number; unit: participants
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 229 | 115
participants | 128 | 14
Statistical Analysis 1: Comparison: Adalimumab/Adalimumab vs Placebo/Adalimumab; Test type: Superiority or Other; p < 0.001, Chi-squared

6. Secondary Outcome: Number of Participants Meeting the ASAS5/6 Response Criteria
Description: as for outcome 5
Time Frame: Week 24
Population: ITT analysis set, missing data imputed by NRI
Measure: Number; unit: participants
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 224 | 113
participants | 150 | 69

7. Secondary Outcome: Number of Participants With ASAS Partial Remission
Description: Participants were classified as having achieved ASAS partial remission if they had a value of less than 20 on a scale from 0 (normal/none) to 100 (most severe) in each of 4 domains: Patient's Global Assessment of Disease Activity; pain as measured by the Total Back Pain visual analog scale (VAS); function as measured by the Bath Ankylosing Spondylitis Functional Index (BASFI); and inflammation (mean of 2 morning stiffness-related Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] scores).
Time Frame: Week 12
Population: ITT analysis set, missing data imputed by NRI
Measure: Number; unit: participants
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 229 | 115
participants | 50 | 4
Statistical Analysis 1: Comparison: Adalimumab/Adalimumab vs Placebo/Adalimumab; Test type: Superiority or Other; p < 0.001, Chi-squared

8. Secondary Outcome: Number of Participants With ASAS Partial Remission
Description: as for outcome 7
Time Frame: Week 24
Population: ITT analysis set, missing data imputed by NRI
Measure: Number; unit: participants
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 224 | 113
participants | 85 | 33

9. Secondary Outcome: Change From Baseline in Patient Global Assessment of Disease Activity
Description: Participants assessed their disease activity during the preceding week using a 100 millimeter (mm) visual analog scale, with responses ranging from no activity (0) to severe activity (100).
Time Frame: Baseline and Week 12
Population: ITT analysis set, missing data imputed by last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 229 | 115
millimeters | -28.8 (24.16) | -11.7 (21.77)
Statistical Analysis 1: Comparison: Adalimumab/Adalimumab vs Placebo/Adalimumab; Test type: Superiority or Other; p < 0.001, ANCOVA

10. Secondary Outcome: Change From Baseline in Patient Global Assessment of Disease Activity
Description: as for outcome 9
Time Frame: Baseline and Week 24
Population: ITT analysis set, missing data imputed by last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 224 | 113
millimeters | -37.8 (24.47) | -35.5 (25.03)

11. Secondary Outcome: Change From Baseline in Total Back Pain Score
Description: Participants assessed their total back pain within the preceding week using a total back pain 100 mm visual analog scale, with responses ranging from no pain (0) to most severe pain (100).
Time Frame: Baseline and Week 12
Population: ITT analysis set, LOCF
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 229 | 115
millimeters | -32.0 (23.55) | -13.7 (22.88)
Statistical Analysis 1: Comparison: Adalimumab/Adalimumab vs Placebo/Adalimumab; Test type: Superiority or Other; p < 0.001, Chi-squared, Corrected

12. Secondary Outcome: Change From Baseline in Total Back Pain Score
Description: as for outcome 11
Time Frame: Baseline and Week 24
Population: ITT analysis set, LOCF
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 224 | 113
millimeters | -42.1 (23.29) | -37.8 (24.20)

13. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) Score
Description: Participants assessed their ability to perform 10 selected activities (e.g., putting on socks or tights without help or aids, bending forward from the waist to pick up a pen from the floor without an aid) during the preceding week. Responses ranged from 0 (easy) to 100 (impossible). The BASFI score is the average of the 10 responses and has a possible minimum value of 0 and a possible maximum value of 100.
Time Frame: Baseline and Week 12
Population: ITT analysis set, LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 229 | 115
units on a scale | -17.5 (20.18) | -4.7 (16.40)
Statistical Analysis 1: Comparison: Adalimumab/Adalimumab vs Placebo/Adalimumab; Test type: Superiority or Other; p < 0.001, ANCOVA

14. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) Score
Description: as for outcome 13
Time Frame: Baseline and Week 24
Population: ITT analysis set, LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 224 | 113
units on a scale | -23.2 (21.03) | -20.9 (21.51)

15. Secondary Outcome: Change From Baseline in Inflammation Score
Description: The Inflammation score is the mean of the 10-cm visual analog scale scores from the 2 morning stiffness-related BASDAI questions: "How would you describe the overall level of morning stiffness you have had from the time you wake up?", with response ranging from none to very severe; and "How long does your morning stiffness last from the time you wake up?", with response ranging from 0 hours to 2 or more hours.
Time Frame: Baseline and Week 12
Population: ITT analysis set, LOCF
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 229 | 115
centimeters | -2.9 (2.01) | -1.5 (2.16)
Statistical Analysis 1: Comparison: Adalimumab/Adalimumab vs Placebo/Adalimumab; Test type: Superiority or Other; p < 0.001, ANCOVA

16. Secondary Outcome: Change From Baseline in Inflammation Score
Description: as for outcome 15
Time Frame: Baseline and Week 24
Population: ITT analysis set, LOCF
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 224 | 113
centimeters | -3.6 (2.21) | -3.6 (2.24)

17. Secondary Outcome: Number of Participants Meeting the Bath Ankylosing Spondyloarthritis Disease Activity Index (BASDAI) BASDAI50 Response Criteria
Description: A BASDAI50 responder had at least a 50% improvement from Baseline in BASDAI score. In the BASDAI, participants use a 10-centimeter visual analog scale to answer 6 questions pertaining to symptoms experienced in the preceding week (e.g., How would you describe the overall level of fatigue/tiredness you have experienced? How long does your morning stiffness last from the time you wake up?) Responses range from "none" to "very severe" or from 0 hours to 2 or more hours for morning stiffness. The score is calculated as 0.2 (Q1 + Q2 + Q3 + Q4 + Q5/2 + Q6/2).
Time Frame: Week 12
Population: ITT analysis set, missing data imputed by NRI
Measure: Number; unit: participants
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 229 | 115
participants | 114 | 19
Statistical Analysis 1: Comparison: Adalimumab/Adalimumab vs Placebo/Adalimumab; Test type: Superiority or Other; p < 0.001, Chi-squared

18. Secondary Outcome: Number of Participants Meeting the Bath Ankylosing Spondyloarthritis Disease Activity Index (BASDAI) BASDAI50 Response Criteria
Description: as for outcome 17
Time Frame: Week 24
Population: ITT analysis set, missing data imputed by NRI
Measure: Number; unit: participants
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 224 | 113
participants | 156 | 71

19. Secondary Outcome: Change From Baseline in High-sensitivity C-Reactive Protein (Hs-CRP)
Description: Elevation of hs-CRP is a nonspecific marker of inflammation. Values above 5 milligrams/liter (mg/L) were considered abnormally high. Decrease in level of hs-CRP indicates reduction in inflammation.
Time Frame: Baseline and Week 12
Population: ITT analysis set, LOCF
Measure: Mean (Standard Deviation); unit: milligrams/liter
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 229 | 115
milligrams/liter | -17.8 (23.76) | -4.2 (21.23)
Statistical Analysis 1: Comparison: Adalimumab/Adalimumab vs Placebo/Adalimumab; Test type: Superiority or Other; p < 0.001, ANCOVA

20. Secondary Outcome: Change From Baseline in High-sensitivity C-Reactive Protein (Hs-CRP)
Description: as for outcome 19
Time Frame: Baseline and Week 24
Population: ITT analysis set, LOCF
Measure: Mean (Standard Deviation); unit: milligrams/liter
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 224 | 113
milligrams/liter | -18.2 (24.27) | -20.1 (30.63)

21. Secondary Outcome: Change From Baseline in 36-item Short Form Questionnaire Version 2 (SF-36v2) Physical Component Summary Score
Description: The SF-36 questionnaire, version 2, consists of 36 general health questions with 2 components, physical and mental. For each component, a transformed summary score is calculated using 8 sub-domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Scores range from 0 to 100. Higher scores indicate a better health state.
Time Frame: Baseline and Week 12
Population: ITT analysis set, observed cases
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 226 | 113
units on a scale | 6.6 (6.43) | 4.0 (6.31)
Statistical Analysis 1: Comparison: Adalimumab/Adalimumab vs Placebo/Adalimumab; Test type: Superiority or Other; p < 0.001, ANCOVA

22. Secondary Outcome: Change From Baseline in 36-item Short Form Questionnaire Version 2 (SF-36v2) Physical Component Summary Score
Description: as for outcome 21
Time Frame: Baseline and Week 24
Population: ITT analysis set, observed cases
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab/Adalimumab | Placebo/Adalimumab
Number analyzed (Participants) | 222 | 110
units on a scale | 8.6 (7.44) | 9.2 (7.25)

ADVERSE EVENTS:
Time Frame: All adverse events reported from the time of first study drug administration until 70 days following discontinuation of study drug administration were collected, for a maximum reporting period of 32 weeks.
Groups:
- Adalimumab (Period 1): Blinded adalimumab from Week 0 to Week 10
- Placebo (Period 1): Blinded placebo from Week 0 to Week 10
- Adalimumab/Adalimumab (Period 2): Open-label adalimumab from Week 12 to Week 22 in participants previously on blinded adalimumab from Week 0 to Week 10
- Placebo/Adalimumab (Period 2): Open-label adalimumab from Week 12 to Week 22 in participants previously on blinded placebo from Week 0 to Week 10
Arm/Group | Adalimumab (Period 1) | Placebo (Period 1) | Adalimumab/Adalimumab (Period 2) | Placebo/Adalimumab (Period 2)
Serious Adverse Events (participants affected / at risk) | 1/229 | 1/115 | 3/224 | 1/113
Other Adverse Events (participants affected / at risk) | 55/229 | 16/115 | 32/224 | 22/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (Period 1) (N=229) | Placebo (Period 1) (N=115) | Adalimumab/Adalimumab (Period 2) (N=224) | Placebo/Adalimumab (Period 2) (N=113)
Hepatitis viral (Infections and infestations) | 0 | 0 | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 1 | 0 | 0 | 0
Peritoneal tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 — Note: One subject had 3 tuberculosis-related adverse events (peritoneal tuberculosis, pulmonary tuberculosis, and tuberculous pleurisy).
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Tuberculosis pleurisy (Infections and infestations) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 — Note: One subject had 3 injury-related adverse events (concussion, contusion, and skin laceration).
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Abortion induced (Surgical and medical procedures) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (Period 1) (N=229) | Placebo (Period 1) (N=115) | Adalimumab/Adalimumab (Period 2) (N=224) | Placebo/Adalimumab (Period 2) (N=113)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Injection site erythema (General disorders) | 4 | 0 | 0 | 1
Injection site swelling (General disorders) | 1 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 4 | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 13 | 9 | 13 | 8
Alanine aminotransferase increased (Investigations) | 26 | 2 | 11 | 13
Aspartate aminotransferase increased (Investigations) | 20 | 1 | 6 | 9
Blood alkaline phosphatase increased (Investigations) | 3 | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 4 | 0
Blood triglycerides increased (Investigations) | 3 | 1 | 2 | 2
Platelet count decreased (Investigations) | 2 | 0 | 4 | 0
White blood cell count decreased (Investigations) | 6 | 2 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.